CLINICAL TRIAL: NCT01908530
Title: Clinical Assessment of a Novel Microprobe Array Continuous Glucose Monitor for Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13SM0639
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Continuous Glucose Monitoring; Microprobes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microprobe Glucose Sensor Phase 1 (Experimental): The microprobe array continuous glucose sensor will be applied to healthy volunteers for 6 hours
  Interventions: Device: Microprobe glucose sensor
- Microprobe Glucose Sensor Phase 2 (Experimental): The microprobe array continuous glucose sensor will be applied to healthy volunteers for 24 hours
  Interventions: Device: Microprobe glucose sensor
- Microprobe Glucose Sensor Phase 3 and 4 (Experimental): The microprobe array continuous glucose sensor will be applied to participants with type 1 diabetes
  Interventions: Device: Microprobe glucose sensor

INTERVENTIONS:
Device: Microprobe glucose sensor — Assessment of safety and accuracy of a novel continuous glucose monitor based on microprobe technology.
  Other Names: Microprobe Array Continuous Glucose Monitor

SUMMARY:
The purpose of the study is to assess the safety and efficacy of the Imperial College Microprobe Array Continuous Glucose Sensor in healthy volunteers and in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
Continuous knowledge of ambient glucose levels will be of benefit to patients with T1DM, especially those with troublesome hypoglycaemia. Existing monitors require skin puncture to access interstitial fluid and sense its glucose content. Despite their clinical benefits, their use is associated with discomfort and their accuracy is questionable in hypoglycaemia. The development of a painless continuous glucose monitor is regarded as the top research priority by patients with diabetes. A novel continuous glucose monitoring device has been developed at Imperial College based on microprobe technology. It consists of a small, wearable patch (~1 cm2), the size of a conventional postage stamp, containing microscopic projections (microprobes) that penetrate only the outermost skin layer. It accesses interstitial fluid to sense its glucose content without stimulating skin nerve fibres or reaching blood vessels within skin layers. The microprobe surface has the consistency of sandpaper. It is pushed into the skin with an applicator allowing it to penetrate through the skin layers and access the interstitial fluid in a minimally invasive manner. The device is disposable and optimum performance will be assessed over five days. The advantages of microprobe technology have been demonstrated in other clinical situations and include painless insertion, absence of bleeding and a low infection risk. The large surface area utilised in our microprobe device has the potential to improve device sensitivity and accuracy. Pre-clinical validation tests have demonstrated the ability of the device to respond accurately to variable glucose concentrations and to penetrate the outermost skin layer without fracture. We aim now to further develop the device through clinical studies in non-diabetic subjects and subjects with type 1 diabetes to allow painless accurate continuous glucose monitoring.

The study will recruit 16 non-diabetic subjects and 20 subjects with type 1 diabetes.

It will be conducted over four phases;

oPhase 1 will assess safety, as a primary outcome, and efficacy, as a secondary outcome, in non-diabetic subjects over six hours in the clinical research facility where the device will be fitted and a cannula inserted for venous sampling every 15 minutes to measure venous blood glucose (YSI). Safety will be assessed with regards to skin inflammation and pain. Efficacy will be assessed in this phase by assessing magnitude of current measured by the microprobe array sensor and comparison of measured ISF glucose concentrations to simultaneous venous blood glucose samples (YSI).

oPhase 2 will also assess safety, as a primary outcome, and efficacy, as a secondary outcome, in non-diabetic subjects over a period of 24 hours. The first six hours in the clinical research facility (same as phase 1), then subject will be allowed to go home with the device to assess safety over that period.

oPhase 3 aims to assess efficacy of the device as a primary outcome and safety as a secondary outcome. This will be in subjects with type 1 diabetes over 24 hours as inpatients. Efficacy will be assessed mechanically (by the ability to penetrate the stratum corneum) and functionally (by the ability to accurately sense ISF glucose). The derived ISF glucose levels will be compared with simultaneous venous glucose samples (YSI) and with a commercially available CGM device (iPro2, Medtronic). Assessment of microprobe penetration of the stratum corneum will be performed using confocal microscopy, optical coherence tomography and in skin biopsies.

oPhase 4 aims to assess efficacy of the device as a primary outcome and safety as a secondary outcome. This will be in subjects with type 1 diabetes over 5 days in ambulatory situation. Efficacy will be assessed by comparing microprobe sensor derived ISF glucose levels against ISF glucose levels measured using a commercially available CGM device (iPro2, Medtronic).

ELIGIBILITY:
For phases 1 and 2:

Inclusion Criteria:

• Adults over 18 years of age

Exclusion Criteria:

* History of upper limb neuropathy or radiculopathy
* History of pre-existing skin condition
* Pregnant or planning pregnancy in next 12 months
* Breastfeeding
* Enrolled in other clinical trials
* uncontrolled concurrent illness
* Have active malignancy or under investigation for malignancy

For phases 3 and 4:

Inclusion Criteria:

* Adults over 18 years of age.
* Diagnosed with Type 1 diabetes for greater than 1 year.
* HbA1c less than or equal to 9.0 % (75 mmol/mol).
* Registered with a General Practitioner.

Exclusion criteria:

* History of diabetic dermopathy or pre-existing skin condition
* History of upper limb neuropathy or radiculopathy
* Pregnant or planning pregnancy in next 12 months
* Breastfeeding
* Enrolled in other clinical trials
* uncontrolled concurrent illness
* physical or visual impairment preventing sensor's use
* Have active malignancy or under investigation for malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Johnston, PhD, FRCP, Principal Investigator — Professor of Diabetes & Endocrinology - Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Laboudi A, Oliver NS, Cass A, Johnston D. Use of microneedle array devices for continuous glucose monitoring: a review. Diabetes Technol Ther. 2013 Jan;15(1):101-15. doi: 10.1089/dia.2012.0188. Epub 2012 Dec 12. PMID 23234256
- [Background] Pickup JC, Freeman SC, Sutton AJ. Glycaemic control in type 1 diabetes during real time continuous glucose monitoring compared with self monitoring of blood glucose: meta-analysis of randomised controlled trials using individual patient data. BMJ. 2011 Jul 7;343:d3805. doi: 10.1136/bmj.d3805. PMID 21737469
- [Background] Battelino T, Phillip M, Bratina N, Nimri R, Oskarsson P, Bolinder J. Effect of continuous glucose monitoring on hypoglycemia in type 1 diabetes. Diabetes Care. 2011 Apr;34(4):795-800. doi: 10.2337/dc10-1989. Epub 2011 Feb 19. PMID 21335621
- [Background] Khanna P, Strom JA, Malone JI, Bhansali S. Microneedle-based automated therapy for diabetes mellitus. J Diabetes Sci Technol. 2008 Nov;2(6):1122-9. doi: 10.1177/193229680800200621. PMID 19885301
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 4 did not go ahead
Groups:
- Microprobe Glucose Sensor Phase 1: The microprobe array continuous glucose sensor applied to healthy volunteers for 6h
- Microprobe Glucose Sensor Phase 2: The microprobe array continuous glucose sensor applied to healthy volunteers for 24 h
- Microprobe Glucose Sensor Phase 3: The microprobe array continuous glucose sensor applied to participants with type 1 diabetes
Period: Overall Study
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Started | 8 | 8 | 10
Completed | 8 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Microprobe Glucose Sensor Phase 1: The microprobe array continuous glucose sensor applied to healthy volunteers for 6 h
- Microprobe Glucose Sensor Phase 2: The microprobe array continuous glucose sensor will be applied to healthy volunteers for 24 h
- Total: Total of all reporting groups
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3 | Total
Number analyzed (Participants) | 8 | 8 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (6.9) | 34.6 (6.9) | 38 (16) | 35.73 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 4 | 4 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 3 | 3 | 9 | 15
  Race: Asian | 2 | 2 | 0 | 4
  Race: European | 3 | 3 | 0 | 6
  Race: Mixed Race | 0 | 0 | 1 | 1
  Race: Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Developed the Skin Inflammation
Description: The study aims to assess safety of the use of microprobe array continuous glucose sensor with regards to skin inflammation.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Number analyzed (Participants) | 8 | 8 | 10
Participants | 0 | 0 | 0

2. Primary Outcome: Difference to the Venous Blood Glucose MARD
Description: Phase 3 of the study aim to assess efficacy of the device in people with type 1 diabetes. This will be done in comparison to venous blood glucose using YSI machine in a controlled environment over 24 hours (phase 3). it was originally planned to then compare this to ISF glucose in ambulatory situation over five days (phase 4) however phase 4 did not go ahead. Measured using mean absolute relative difference with respect to venous blood glucose
Time Frame: 24 hours
Population: Only for Phase 3 arm
Measure: Number; unit: percentage
Groups:
- Microprobe Glucose Sensor Phase 2: The microprobe array continuous glucose sensor applied to healthy volunteers for 24h
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Number analyzed (Participants) | 0 | 0 | 10
percentage |  |  | 4

3. Secondary Outcome: Pain Score
Description: The study aims to assess safety of the device with regards to pain degree in comparison to venflon insertion and insertion of an existing continuous glucose monitor (Medtronic iPro2 CGM system, Northridge, California). This will be done at each phase of the four study phases.
Time Frame: 24 hours
Population: Data not collected
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participant Developed Skin Penetration
Description: This done using Optical Coherence Tomography and Confocal Microscopy. Measure = variation in penetration depth of microprobe needles over 24 hours
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Number analyzed (Participants) | 8 | 8 | 10
Participants | 0 | 0 | 0

5. Secondary Outcome: Detectable Signal
Description: This is a secondary outcome for phases 1 & 2.
Time Frame: 24 hours
Population: Data not collected
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Correlation With Venous Blood Glucose
Description: This is a secondary outcome for phases 1 and 2. It is a primary outcome for phase 3. Using MARD.
Time Frame: 24 hours
Population: Data not collected
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Acceptability Questionnaire
Description: This is a secondary outcome for phases 3 and 4.
Time Frame: 24 hours
Population: Data not collected
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Microprobe Glucose Sensor Phase 1 | Microprobe Glucose Sensor Phase 2 | Microprobe Glucose Sensor Phase 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT01908530/Prot_000.pdf